CLINICAL TRIAL: NCT00209664
Title: Phase II Study of Oral S-1 Plus Irinotecan in Patients With Advanced Gastric Cancer: Hokkaido Gastrointestinal Cancer Study Group HGCSG0303
Brief Title: Phase II Study of Oral S-1 Plus Irinotecan in Patients With Advanced Gastric Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0303
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2004-01

CONDITIONS: Gastric Cancer
Keywords: Irinotecan, S-1, Phase II, gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; S 1 (combination)

INTERVENTIONS:
Drug: irinotecan
Drug: S-1

SUMMARY:
To assess the usefulness of irinotecan plus S-1 therapy based on the antitumor effect and survival period. by performing a phase II study of this combination in patients with inoperable or with postoperative gastric cancer

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase II clinical trial is conducted on patients with histological stage IV gastric cancer given irinotecan plus S-1. The usefulness of this regimens as 1st line therapy for gastric cancer was evaluated by the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

・ Eligibility criteria

1. Histological diagnosis of gastric adenocarcinoma.
2. Measurable or assessable lesions.
3. Age: 18 ~ 75 years.
4. Performance Status (ECOG): 0 ~ 2.
5. No prior chemotherapy or only one regimen of previous chemotherapy (with a washout period >4 weeks after the final day of the previous therapy). Adjuvant chemotherapy is not defined as previous therapy.
6. No history of treatment with CPT-11 or S-1.
7. No history of radiotherapy to the abdomen.
8. Oral intake of S-1 is possible.
9. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and 12,000/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5times the upper limit of normal (excluding liver metastasis). T-Bil 2.0mg/dl. Creatinine <1.5 mg/dl (but if it is 1.0 ~ 1.5 mg/dl, the dose of S-1 can be decreased according to the dose reduction criteria to allow registration in the trial). Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes). (10) Predicted survival for >3 months.

(11) Able to give written informed consent

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2008-12

PRIMARY OUTCOMES:
objective tumor response

SECONDARY OUTCOMES:
Response duration, time to progression, median survival time, and safety will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshito Komatsu, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan